CLINICAL TRIAL: NCT01319032
Title: Genetic Polymorphism and Israeli Top-level Swimmers' Performance and Expertise
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Wingate Institute (Other)
Responsible Party: Eias Kassem, MD, Hillel Yaffe Medical Center
Other Study IDs: 0013-11-HYMC
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2011-03-21 (Estimated); Status verified 2011-03

CONDITIONS: Genetic Polymorphism Connected to Top-level Swimmers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- I. Top-level swimmers
  Interventions: Other: Extraction of whole blood
- II. Control: Other swimmers
  Interventions: Other: Extraction of whole blood

INTERVENTIONS:
Other: Extraction of whole blood — Extraction of DNA from whole blood

SUMMARY:
In a study conducted in our laboratory few years ago, we genotyped 22 genes in 2 athletic groups (endurance and sprinters) and in age and gender matched nonathletic controls. Few of these genes were found to be associated with athletic performance and area of specificity. Since then a few more genes have been found that are related to athletic performance, and we intend to study various genes related to 3 genetic cascade: genes associated with body fluid balance and homeostasis, genes associated with muscle strength, and genes associated with bioenergy. The results of this study compared with athletic level will provide deeper insight into the genetic mechanisms involved in performance.

ELIGIBILITY:
Inclusion Criteria:

* Top-level swimmers
* Other swimmers

Exclusion Criteria:

* All others

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Swimmers training at the Wingate Institute
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genes associated with swimming performance | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate Institute, Netanya, Israel

REFERENCES:
- [Derived] Ben-Zaken S, Eliakim A, Nemet D, Rabinovich M, Kassem E, Meckel Y. ACTN3 Polymorphism: Comparison Between Elite Swimmers and Runners. Sports Med Open. 2015;1(1):13. doi: 10.1186/s40798-015-0023-y. Epub 2015 Jun 14. PMID 26284168